CLINICAL TRIAL: NCT01179230
Title: A Prospective Comparison of Gated, Rest/Stress Rubidium-82 Position Emission Computed Tomography (PET) vs. Gated, Rest / Stress Technetium 99-m SPECT
Brief Title: Rubidium-82 Position Emission Computed Tomography (PET) Versus Gated, Rest / Stress Technetium 99-m SPECT
Acronym: PETvsSPECT
Status: Completed | Type: Observational
Sponsor: Hartford Hospital (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HELL001671HE
Record Dates: First submitted 2010-06-08; First posted 2010-08-11 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Heart Disease
Keywords: CAD; chest pain; acute coronary syndrome; Myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Heart Diseases; Chest Pain; Acute Coronary Syndrome | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET SPECT: Subjects will have both types of imaging performed, PET and SPECT
  Interventions: Other: SPECT imaging; Other: PET imaging

INTERVENTIONS:
Other: SPECT imaging — Dipyridamole stress testing 0.57 mg/kg
  Other Names: Pharmacological stress testing; Myocardial perfusion imaging; Persantine stress test
Other: PET imaging — Dipyridamole stress test 0.57 mg/kg with Rubidium PET images
  Other Names: PET perfusion images; Rb-92; PET persantine stress test

SUMMARY:
Many stress tests being done today have two parts, the stress test and the pictures of your heart. The investigators are comparing a newer technique to obtain the pictures (PET imaging) to the standard method (SPECT imaging). However, it is not known if the new test is better than the old test. It is important to have a standard to compare these tests to, and that is why people who will be getting a cardiac catheterization are being asked to participate. The information about your arteries from the cardiac catheterization will be used to judge which stress test is better. The investigators hypothesize that the newer method (PET imaging) will be more accurate than the old method (SPECT) in detecting heart disease.

DETAILED DESCRIPTION:
A SPECT rest image will be obtained using a technetium based isotope. On a separate day, a Rubidium rest PET image will be obtained prior to a Dipyridamole stress test. Subjects will receive both Rubidium and technetium isotopes following the Dipyridamole stress, and will undergo first PET imaging and later SPECT imaging following the stress test. Patients will then go for cardiac catheterization as clinically ordered by their physician.

ELIGIBILITY:
Inclusion Criteria:

* referred for clinical cardiac catheterization

Exclusion Criteria:

* previous CABG
* previous MI
* Asthma or obstructive airway disease
* Intolerance to Dipyridamole
* Moderate to severe valvular disease
* Cardiomyopathy - (ejection fraction less than 45%)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate to high likelihood of CAD referred for cardiac catheterization, either on outpatient or inpatient basis
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2005-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Disease | 30 days

SECONDARY OUTCOMES:
Myocardial Ischemia | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary V. Heller, M.D., Ph.D., Principal Investigator — Hartford Hospital
Locations (5):
- United States (5):
  - The Heart Center, PC, Huntsville, Alabama
  - Hartford Hospital, Hartford, Connecticut
  - Cardiovascular Imaging Technologies, LLC, Kansas City, Missouri
  - Sanford Health Clinical Research, Fargo, North Dakota
  - Ohio Health Research Institute, Columbus, Ohio

REFERENCES:
- [Background] Bateman TM, Heller GV, McGhie AI, Friedman JD, Case JA, Bryngelson JR, Hertenstein GK, Moutray KL, Reid K, Cullom SJ. Diagnostic accuracy of rest/stress ECG-gated Rb-82 myocardial perfusion PET: comparison with ECG-gated Tc-99m sestamibi SPECT. J Nucl Cardiol. 2006 Jan-Feb;13(1):24-33. doi: 10.1016/j.nuclcard.2005.12.004. PMID 16464714
- [Background] Freedman N, Schechter D, Klein M, Marciano R, Rozenman Y, Chisin R. SPECT attenuation artifacts in normal and overweight persons: insights from a retrospective comparison of Rb-82 positron emission tomography and TI-201 SPECT myocardial perfusion imaging. Clin Nucl Med. 2000 Dec;25(12):1019-23. doi: 10.1097/00003072-200012000-00014. PMID 11129138
- [Background] Stewart RE, Schwaiger M, Molina E, Popma J, Gacioch GM, Kalus M, Squicciarini S, al-Aouar ZR, Schork A, Kuhl DE. Comparison of rubidium-82 positron emission tomography and thallium-201 SPECT imaging for detection of coronary artery disease. Am J Cardiol. 1991 Jun 15;67(16):1303-10. doi: 10.1016/0002-9149(91)90456-u. PMID 2042560
- [Background] Go RT, Marwick TH, MacIntyre WJ, Saha GB, Neumann DR, Underwood DA, Simpfendorfer CC. A prospective comparison of rubidium-82 PET and thallium-201 SPECT myocardial perfusion imaging utilizing a single dipyridamole stress in the diagnosis of coronary artery disease. J Nucl Med. 1990 Dec;31(12):1899-905. PMID 2266384